CLINICAL TRIAL: NCT06732167
Title: Prospective, Randomized, Controlled, Multicenter Study on the Performance and Safety of Lyoplant® in Guided Bone Regeneration (GBR) in Oral Surgery
Brief Title: Performance and Safety of Lyoplant® in Guided Bone Regeneration (GBR) in Oral Surgery
Acronym: LyOral
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-2014
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Bone Regeneration
Keywords: collagen barrier membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyoplant® (Experimental)
  Interventions: Procedure: GBR Lyoplant
- Bio-Gide® (Active Comparator)
  Interventions: Procedure: GBR Bio-Gide

INTERVENTIONS:
Procedure: GBR Lyoplant — GBR surgical procedure with simultaneous implant placement including membrane placement
  Arms: Lyoplant®
Procedure: GBR Bio-Gide — GBR surgical procedure with simultaneous implant placement including membrane placement
  Arms: Bio-Gide®

SUMMARY:
Guided Bone Regeneration (GBR) is a well-established surgical technique that employs barrier membranes to ensure the stability of bone augmentation material while preventing the infiltration of soft tissue, thereby facilitating new bone formation.

The primary objective of this randomized controlled trial is to assess the performance and safety of the Lyoplant® collagen membrane as a barrier membrane in GBR for patients undergoing dental implant surgery. Additionally, the study aims to compare the Lyoplant® membrane with the Bio-Gide® collagen membrane, with the goal of demonstrating the non-inferiority of the Lyoplant® membrane in terms of radiographically measured bone gain compared to the comparator.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to give a voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the Informed Consent Form (ICF).
* Patients with the capacity to consent for themselves.
* Patients in need of an implant with a simultaneous GBR procedure.
* Presence of buccal bony dehiscence with a vertical defect height (VDH) ≥ 1 mm and ≤ 6 mm after implant placing.
* The tooth at the implant site must have been extracted or lost at least 8 weeks before the date of bone augmentation (volumetrically healed site).

Exclusion Criteria:

* Patients < 18 years.
* Currently pregnant or breastfeeding women.
* Major systemic diseases (e.g. recent myocardial infarction, cerebrovascular accident or valvular prosthesis surgery, a poorly stabilized diabetes mellitus, severe hypertension, severe peripheral artery occlusive disease, malignancies, autoimmune diseases, or kidney diseases, untreated or uncontrolled periodontal disease, uncontrolled drug or alcohol abuse, uncontrolled psychiatric disorders).
* Acute infectious diseases.
* Immunocompromised patients.
* Serious disturbances of bone metabolism and/or serious bone diseases of endocrine etiology.
* Medical conditions requiring prolonged use (> 6 months) of steroids and/or ongoing treatment with gluco- and mineralocorticoids and with agents affecting calcium metabolism (e.g. calcitonin), and/or anticoagulative therapy.
* Previous or current use of antiresorptive drugs (ARDs) (e.g. bisphosphonates, selective estrogen receptor modulators (SERMs), denosumab, hormone replacement therapy and calcitonin).
* Previous oral / maxillofacial radiotherapy.
* Heavy smoker (>10 cigarettes/day). In the case of vapors with nicotine, the use of >300 puff vapors (equivalent to 10 cigarettes/day) are not allowed.
* Health conditions, which do not permit the surgical treatment.
* Use of the Investigational Device / Comparator in infected areas.
* Known foreign body sensitivity to implant materials.
* Simultaneous participation in another interventional clinical trial (drugs or medical devices studies) if it could impact the result of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Gain of horizontal bone thickness at the augmented site | At Visit 5: 5 months after GBR intervention
  At Visit 2 (V2) and Visit 5 (V5) a Cone Beam Computed Tomography (CBCT) is taken. CBCTs are compared and horizontal bone dimensions at augmented site are measured at four levels (at implant shoulder, 2 mm, 4 mm, and 6 mm from the implant shoulder).

SECONDARY OUTCOMES:
Number of side effects | At each follow-up visit: V3 (after 7-14 days), V4 (after 1 month ± 7 days) and V5 (after 5 months ± 2 weeks)
  Side effects to be assessed are:
  * Wound infection
  * Wound dehiscence
  * Membrane exposure
  * Flap sloughing
  * Foreign body reaction
  * Abscess/pus formation
  * Redness/swelling
Number of safety endpoints | At each follow-up visit: V3 (after 7-14 days), V4 (after 1 month ± 7 days) and V5 (after 5 months ± 2 weeks)
  Safety endpoints to be assessed are:
  * Device related adverse events (adverse device effects (ADE)
  * Seriousness of device related adverse events (serious adverse device effect (SADE))
  * Device deficiency (DD)
Membrane usability | At V2 (surgery): directly after GBR intervention
  The usability of Lyoplant® and Bio-Gide® membranes will be evaluated by completing a survey regarding the handling of these membranes (measured on a 5-point Likert scale) by the Investigator.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Odontològic Universitat de Barcelona, Campus Ciències de la Salut de Bellvitge, Barcelona, Catalonia
  - Clínica Universitaria d.Odontologia de la Universitat Internacional de Catalunya, Sant Cugat Del Vallés, Catalonia